CLINICAL TRIAL: NCT06262672
Title: The Relationship Between Healthy Lifestyle Behaviors, Sleep Quality, and Body Weight in University Students During the COVID-19 Epidemic Process
Brief Title: Evaluation of Some Parameters in University Students During the COVİD-19 Epidemic Process
Status: Completed | Type: Observational
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Fulya Demirhan, Research Assistant, Kırklareli University
Other Study IDs: PR0319R01
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Health Behavior; Sleep; Body Weight
MeSH Terms: conditions — Health Behavior; Body Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation form — This form is a form of demographic information, questions that question the habits of COVİD-19 era, and evaluation scales.

SUMMARY:
The physical and mental effects of the COVID-19 pandemic have been examined by many researchers, but this study aims to evaluate in every aspect how university students who had to receive education with the distance education model due to the pandemic went through this process. Data regarding people's positive and negative habits from anthropometric characteristics and sleep quality, which is one of the sub-dimensions of healthy lifestyle behaviors, were evaluated, and the relationship between these parameters was examined in detail.

DETAILED DESCRIPTION:
This study focuses on distance education, remote working, etc. during the pandemic period. It is compatible with the findings of studies on the subject and reveals that the nutrition and physical activity sub-parameters of the healthy lifestyle behaviors scale are related to anthropometric characteristics and sleep quality. Considering that the online working model has become widespread, from this perspective, for future studies, the effects of behavioral change strategies on individuals' sleep quality and anthropometric values can be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Students who are registered to Kırklareli University Faculty of Health Sciences and aged 18 years and older who agreed to participate in the study
* Those who are capable of filling out surveys online
* Those with internet access
* With the fully answered to the questionnaire and scale questions

Exclusion Criteria:

* Students who are not registered to Kırklareli University Faculty of Health Sciences

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students registered to Kırklareli University Faculty of Health Sciences and attending distance education due to COVID-19 pandema
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Health Promotion Life-Style Profile (HPLP-II) | Students who filled the survey between 20/11/2021 with 20/05/2021
  The scale measures health-promoting behaviors in relation to an individual's healthy lifestyle. The scale consists of a total of 52 items and has six sub-factors. The subgroups are spiritual development, health responsibility, physical activity, nutrition, interpersonal relationships, and stress management.
Pittsburgh Sleep Quality Index (PSQI) | Students who filled the survey between 20/11/2021 with 20/05/2021
  PSQI, which evaluates the individual's sleep quality in the last month, contains a total of 24 questions. 19 of these are self-reported questions and are answered by the patient himself.
Anthropometric Measurements | Students who filled the survey between 20/11/2021 with 20/05/2021
  Body weights (kg) and height lengths (cm) were taken as anthropometric measurements of individuals, and body mass indexes (BMI) were calculated. WHO classification was used in the evaluation of BMI. According to this classification, the BMI is less than 18.5 kg/m2, weak, 18.5-24.9 kg/m2 are normal, 25.0-29.9 kg/m2 are classified as slightly fat, and over 30 kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Merve PEHLIVAN, Assoc. prof., Principal Investigator — Trakya University
Locations (1):
- Kirklareli University, Kırklareli, Kayalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided